CLINICAL TRIAL: NCT07389343
Title: Immediate Effect of a Semirigid Foot Insole on Radiological Foot Angles in Flexible Pes Planus
Brief Title: Effect of a Semirigid Foot Insole in Flexible Pes Planus
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fatma El Zahraa (Other)
Responsible Party: Sponsor-Investigator, Fatma El Zahraa, lecturer assistant at faculty of physical therapy-Ahram Canadian University AND PHD candidate at Faculty of physical therapy, Cairo University
Organization: Cairo University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Fatma-PhD
Record Dates: First submitted 2026-01-23; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Flexible Flatfoot or Pes Planus
Keywords: "Foot insole" and "Flexible flatfoot" and "radiological foot angles"
MeSH Terms: conditions — Flatfoot | interventions — Foot Orthoses

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Semirigid foot insole (Experimental): A semi-rigidly designed foot insole will be used to investigate the correction provided for flat-foot angles.
  Interventions: Other: Foot Insole

INTERVENTIONS:
Other: Foot Insole — Designed Semirigid foot insole

SUMMARY:
The goal of this clinical trial is to investigate the effect of a semirigid foot insole on radiological angle correction in people with asymptomatic flexible flat feet. The X-ray will be performed while standing barefoot one time and the other while standing on the insole from 2 views.

DETAILED DESCRIPTION:
This study will be conducted on 30 male and female subjects with flexible pes planus. Clinical diagnosis for flexible pes planus will be made through the navicular drop test (NDT) and the Foot Posture Index (FPI). The study included asymptomatic people with flexible pes planus. If the pain is greater than 3 out of 10 on the numeric pain rating scale in the last 3 months, aged 18-35, and BMI max 29.9 kg/cm². The subjects will be excluded if they have osteoarthritis of the joints of the foot (excluded by x-ray), foot deformities (e.g., hallux valgus), old fractures of the foot, previous injuries to the ankle, or previous surgeries to the lower limb. Calcaneal Spur, Foot and Ankle Ligament Tear, Systemic diseases such as rheumatoid arthritis (gouty arthritis, an autoimmune disease) and neurological diseases. The X-ray is the gold standard for assessment of adult-acquired flat foot deformity. Two views are used: anteroposterior (AP) and lateral views. A ruler and protractor will be used for manual measurements of X-ray foot. The subject will stand barefoot, and a weight-bearing X-ray will be taken from lateral and AP views once, without an insole, and another photo will be taken with an insole. The subject will stand barefoot, and a weight-bearing X-ray will be taken from lateral and AP views once, without an insole, and another photo will be taken with an insole.

The angles will be measured:

The gathered angles aim to evaluate the alignment of the foot's three arches. In the lateral view, the following angles will be measured and evaluated with without the insole: the lateral talo-1st metatarsal angle, the calcaneal inclination angle, the angle of Hibbs, the calcaneal-5th metatarsal angle, and the navicular height.

In the AP view, the following angles will be measured and evaluated with without the insole: The lateral talo-1st metatarsal angle, Talo-2nd metatarsal angle, The talocalcaneal angle, Talonavicular coverage angle and First-fifth metatarsal angle

ELIGIBILITY:
Inclusion Criteria:

1. Asymptomatic people with flexible pes planus. If the pain is greater than 3 out of 10 on the visual analog scale in the last 3 months, the patient is considered to have symptomatic flat feet (Mahdiyar et al., 2021).
2. Aged 18-35.
3. BMI max 29.9 kg/cm².

Exclusion Criteria:

1. Osteoarthritis of the joints of the foot (excluded by x-ray).
2. Foot Deformities (e.g. Hallux Valgus)
3. Old fractures of the foot.
4. Previous injuries to the ankle.
5. Previous surgeries to the lower limb. 6. Calcaneal Spur. 7. Foot and ankle ligaments tear.

8- Systemic diseases such as rheumatoid arthritis. (Gouty arthritis, autoimmune disease) 9. Neurological diseases.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08-27 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Radiological foot angles | Immediately after the insole insertion. The radiology will be taken one time barefoot and second time with the insole insertion, and the researcher will measure the foot angles pre- and post-insole to measure the correction.
  In the lateral view,the lateral talo-1st metatarsal angle, the calcaneal inclination angle, the angle of Hibbs, the calcaneal-5th metatarsal angle, and the navicular height.
  In the AP view,The lateral talo-1st metatarsal angle, Talo-2nd metatarsal angle, The talocalcaneal angle, Talonavicular coverage angle and First-fifth metatarsal angle

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Elzahraa A ElBayomi, MSc degree, Principal Investigator — Cairo University
Locations (1):
- October 6 University Hospital, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No
Obtaining the patient privacy, however the data will be available with the original author uopn request